CLINICAL TRIAL: NCT07171424
Title: Moving Beyond p-Values: Minimal Clinically Important Difference for Overactive Bladder Questionnaire - Version 8 and International Consultation on Incontinence Questionnaire - Short Form in Patients With Overactive Bladder Syndrome
Brief Title: Moving Beyond p-Values: MCID for OAB-V8 8 and ICIQ-SF in Patients With OAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCID-2
Record Dates: First submitted 2025-09-06; First posted 2025-09-12 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Overactive Bladder Syndrome
Keywords: overactive bladder; minimal clinically important difference; urinary incontinence; quality of life; ROC curve
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: In this prospective study, one treatment group was formed to receive behavioral therapy and transcutaneous posterior tibial nerve stimulation (TPTNS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Behavioral therapy and transcutaneous posterior tibial nerve stimulation (Experimental): Patients with OAB will receive behavioral therapy and TPTNS one day a week for 12 weeks as previously recommended.
  Interventions: Other: Behavioral therapy and transcutaneous posterior tibial nerve stimulation

INTERVENTIONS:
Other: Behavioral therapy and transcutaneous posterior tibial nerve stimulation — Behavioral therapy included appropriate fluid intake, bladder training, habit training, pelvic floor muscle exercises (Kegel exercises), prompted voiding, and scheduled voiding. TPTNS will be applied in a biphasic square waveform with a frequency of 20 Hz and 200 cycles/sec in 30-minute sessions. The current intensity will be varied between 0.5-20 mA according to the patient's pain threshold.

SUMMARY:
The goal of this study was to determine the Minimal Clinically Important Difference (MCID) for the Overactive Bladder Questionnaire-Version 8 (OAB-V8) and the International Consultation on Incontinence Questionnaire- Short Form (ICIQ-SF) in people with Overactive Bladder Syndrome (OAB).

DETAILED DESCRIPTION:
104 patients with OAB will receive common behavioral therapy and transcutaneous posterior tibial nerve stimulation (TPTNS) for 12 weeks. OAB-related symptoms and quality of life (QoL) will be assessed with the OAB-V8 and ICIQ-SF baseline and post-intervention. The receiver operating characteristic (ROC) analysis and the Gamma coefficient will be employed to determine sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with urge and mixed urinary incontinence symptoms or with OAB symptoms only (no history of urinary incontinence),
* women over 18 years of age.

Exclusion Criteria:

* patients who did not give consent to participate in the study,
* not understanding the instructions given by the researcher,
* pregnancy or planning a pregnancy in the near future,
* urinary tract infection or kidney stones,
* pelvic organ prolapse of grade II or higher,
* stress-type urinary incontinence,
* neurogenic bladder,
* use of a pacemaker,
* epilepsy,
* peripheral neuropathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women with an overactive bladder will be included.
Enrollment: 104 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Questionnaire-Version 8 (OAB-V8) | Baseline
  On this scale, which ranges from 0 to 40 points, higher scores are associated with greater symptom severity.
Overactive Bladder Questionnaire-Version 8 (OAB-V8) | After the 12-week intervention
  On this scale, which ranges from 0 to 40 points, higher scores are associated with greater symptom severity.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire- Short Form (ICIQ-SF) | Baseline
  The total score of the scale ranges from 0 to 21, with higher scores indicating more severe symptoms. It measures the frequency, severity, and impact of OAB through three main questions. An additional open-ended question allows patients to describe their symptoms.
International Consultation on Incontinence Questionnaire- Short Form (ICIQ-SF) | After the 12-week intervention
  The total score of the scale ranges from 0 to 21, with higher scores indicating more severe symptoms. It measures the frequency, severity, and impact of OAB through three main questions. An additional open-ended question allows patients to describe their symptoms.

OTHER OUTCOMES:
Global Rating Change (GRC) | After the 12-week intervention
  The GRC comprised seven responses, ranging from 1 to 5, indicating "very much better," "slightly better," "no change," "slightly worse," and "very much worse," respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, Principal Investigator — Artvin Coruh University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiengthong K, Bunyavejchevin S. Efficacy of Erbium YAG laser treatment in overactive bladder syndrome: a randomized controlled trial. Menopause. 2023 Apr 1;30(4):414-420. doi: 10.1097/GME.0000000000002159. Epub 2023 Feb 27. PMID 36854167
- [Background] Reynolds WS, Fowke J, Dmochowski R. The Burden of Overactive Bladder on US Public Health. Curr Bladder Dysfunct Rep. 2016 Mar;11(1):8-13. doi: 10.1007/s11884-016-0344-9. Epub 2016 Jan 23. PMID 27057265
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Yang DY, Zhao LN, Qiu MX. Treatment for overactive bladder: A meta-analysis of transcutaneous tibial nerve stimulation versus percutaneous tibial nerve stimulation. Medicine (Baltimore). 2021 May 21;100(20):e25941. doi: 10.1097/MD.0000000000025941. PMID 34011072
- [Background] Abrams P, Smith AP, Cotterill N. The impact of urinary incontinence on health-related quality of life (HRQoL) in a real-world population of women aged 45-60 years: results from a survey in France, Germany, the UK and the USA. BJU Int. 2015 Jan;115(1):143-52. doi: 10.1111/bju.12852. Epub 2014 Aug 16. PMID 24958472
- [Background] Coyne KS, Zyczynski T, Margolis MK, Elinoff V, Roberts RG. Validation of an overactive bladder awareness tool for use in primary care settings. Adv Ther. 2005 Jul-Aug;22(4):381-94. doi: 10.1007/BF02850085. PMID 16418145
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Husted JA, Cook RJ, Farewell VT, Gladman DD. Methods for assessing responsiveness: a critical review and recommendations. J Clin Epidemiol. 2000 May;53(5):459-68. doi: 10.1016/s0895-4356(99)00206-1. PMID 10812317
- [Background] Frawley H, Shelly B, Morin M, Bernard S, Bo K, Digesu GA, Dickinson T, Goonewardene S, McClurg D, Rahnama'i MS, Schizas A, Slieker-Ten Hove M, Takahashi S, Voelkl Guevara J. An International Continence Society (ICS) report on the terminology for pelvic floor muscle assessment. Neurourol Urodyn. 2021 Jun;40(5):1217-1260. doi: 10.1002/nau.24658. Epub 2021 Apr 12. PMID 33844342
- [Background] Hu JS, Pierre EF. Urinary Incontinence in Women: Evaluation and Management. Am Fam Physician. 2019 Sep 15;100(6):339-348. PMID 31524367
- [Background] Ramirez-Garcia I, Blanco-Ratto L, Kauffmann S, Carralero-Martinez A, Sanchez E. Efficacy of transcutaneous stimulation of the posterior tibial nerve compared to percutaneous stimulation in idiopathic overactive bladder syndrome: Randomized control trial. Neurourol Urodyn. 2019 Jan;38(1):261-268. doi: 10.1002/nau.23843. Epub 2018 Oct 12. PMID 30311692
- [Background] Greco NJ, Anderson AF, Mann BJ, Cole BJ, Farr J, Nissen CW, Irrgang JJ. Responsiveness of the International Knee Documentation Committee Subjective Knee Form in comparison to the Western Ontario and McMaster Universities Osteoarthritis Index, modified Cincinnati Knee Rating System, and Short Form 36 in patients with focal articular cartilage defects. Am J Sports Med. 2010 May;38(5):891-902. doi: 10.1177/0363546509354163. Epub 2009 Dec 31. PMID 20044494
- [Background] Lehman LA, Velozo CA. Ability to detect change in patient function: responsiveness designs and methods of calculation. J Hand Ther. 2010 Oct-Dec;23(4):361-70; quiz 371. doi: 10.1016/j.jht.2010.05.003. Epub 2010 Jul 17. PMID 20638823